CLINICAL TRIAL: NCT02547051
Title: Dietary Factors and Disfluency. A Look Into Causes and Variations in Severity of Disfluency in Regards to Vocal Cord Tension.
Brief Title: Dietary Factors and Disfluency: A Look Into Food Allergies and Other Environmental Triggers Associated With Variations in Severity of Vocal Cord Tension.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The R2 Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2001AA
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Vocal Cord Tension; Dysfluency Developmental
MeSH Terms: interventions — Elimination Diets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food allergy and vocal cord tension (Experimental): To determine if dietary allergen responses and frequency and severity of vocal cord tension.
  Interventions: Other: Food Allergy Testing and Elimination Diet

INTERVENTIONS:
Other: Food Allergy Testing and Elimination Diet — Food allergy testing and elimination diet

SUMMARY:
The purpose of this study is to see whether participants with persistent developmental disfluency who report fluctuational disfluency due to vocal cord tension on a day to day basis of can achieve a more normalized fluency by identifying dietary allergen responses and subsequently eliminating these dietary triggers from their daily consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients reporting persistent developmental disfluency.

Exclusion Criteria:

* Patients reporting no changes in disfluency severity or frequency

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Dietary Factors and Disfluency: Variations in Severity of Vocal Cord tension | 1 Year
  Initial fluency samples are taken prior to treatment protocol of study.
  Food sensitivity panel will be assessed for potential allergans. Allergan responses are graded from 0 being no response to food allergen to 3 being the strongest response and subsequent removal of sensitive allergan from diet. Speech sample and disfluency severity will be evaluated qualitatively again via the SSI-3 on repeat office visit at fixed interval scale. Erickson S-24 repeated at end of study and final conclusions made.

CONTACTS AND LOCATIONS:
Locations (1):
- R2 Institute, Houston, Texas, United States